CLINICAL TRIAL: NCT01581086
Title: Identify and Characterize Populations at Risk for Developing Pulmonary Arterial Hypertension (PAH)
Brief Title: Vascular Subphenotypes of Lung Disease in HIV & COPD
Acronym: VAST
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: VAST11060550
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2016-05

CONDITIONS: Pulmonary Artery Hypertension
Keywords: HIV; COPD; Pulmonary disease
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is looking for high blood pressure in the lungs (Pulmonary artery hypertension PAH) in HIV and COPD patients.

DETAILED DESCRIPTION:
The goal of the project is to identify and characterize populations at risk for developing pulmonary arterial hypertension (PAH). The project will establish a PAH subphenotype core cohort (CORE) to evaluate mechanistic pathways and test novel therapeutic agents. This core cohort serves as a resource for the Translational Program Project grant, Vascular Subphenotypes of Lung Disease (Mark Gladwin, PI). In order to construct the CORE, we have chosen to recruit COPD and HIV patients, two populations with advanced lung and systemic diseases that are enriched for PAH. We have selected these as prototypic conditions because: A) both COPD patients and HIV-infected patients develop PAH at a rate significantly greater than the general population, B) morbidity and mortality are greatly increased in dually-affected persons, C) mechanisms responsible for development of the PAH "subphenotype" are not well-understood, D) clinical and genetic characteristics of the subgroup with PAH are not known, and E) effects of PAH therapies in subphenotypes are incompletely studied. There is also some overlap between COPD and HIV, with HIV-infected patients having accelerated COPD even with effective antiretroviral therapy. Participants with COPD, HIV, or HIV-uninfected controls will be recruited to the study based on entry criteria of elevated N-terminal pro-brain natriuretic peptide (NT-proBNP) and/or an abnormal echocardiogram. These subjects will then undergo a 6-minute walk test, blood collection, questionnaire, medical record review, and echocardiography (if not previously performed). Selected subjects will then be recruited to undergo right heart catheterization. The goals of the study are to establish a pulmonary hypertension cohort for translational investigations, to determine the utility of NT-proBNP as a biomarker of PAH, to determine clinical characteristics and relationship of lung function to PAH in COPD and HIV, and to establish a biorepository for mechanistic studies of PAH phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female 18-80 years of age.
* Subject has been previously enrolled in PACT/MAC/ECRC study.
* Must have recent ProBNP test >120pg/ml or abnormal echocardiogram (right ventricular systolic pressure >or=40mmHg) without evidence of left sided heart failure.

Exclusion Criteria:

* Previous diagnosis of congenital heart failure.
* If evidence of Left ventricular systolic or diastolic dysfunction, echo will be reviewed by the PI on a case by case basis.
* Creatine clearance <60ml/min per 1.73 m2.
* Undiagnosed chest pain or myocardial infarction, stroke or cardiovascular event within 3 months.
* Pregnancy.
* Subjects receiving chronic anticoagulant.
* Inability to complete the 6 minute walk test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pitt mens Study(MACS).
  University of Pittsburgh HIV Clinic(PACT).
  Emphysema COPD Research Center Research Registry(ECRC).
  University of Pittsburgh Medical center pulmonary hypertension clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
elevated NT-proBNP as a biomarker | 3 years
  establish a pulmonary hypertension cohort for translational investigations, to determine the utility of NT-proBNP as a biomarker of PAH

CONTACTS AND LOCATIONS:
Overall Officials: Michael Risbano, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States